CLINICAL TRIAL: NCT00054262
Title: A Phase II Study Of Intravenous T900607-Sodium In Subjects With Chemotherapy-Naive Unresectable Hepatocellular Carcinoma
Brief Title: T900607 in Treating Patients With Unresectable Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals Seidman Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: TULA-TULI-2202; CWRU-100211; CDR0000270198 (Registry Identifier: PDQ (Physician Data Query)); TULA-T-607-004
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2010-09

CONDITIONS: Liver Cancer
Keywords: localized unresectable adult primary liver cancer; advanced adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — T 900607

INTERVENTIONS:
Drug: T900607

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of T900607 in treating patients who have unresectable liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete and partial response rates of patients with chemotherapy-naïve unresectable hepatocellular carcinoma treated with T900607.
* Determine the efficacy of this drug, in terms of duration of response and time to disease progression, in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Determine the safety profile of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive T900607 IV over 1 hour once weekly. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 20-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed unresectable hepatocellular carcinoma (HCC)
* Bidimensionally measurable disease defined as at least 1 lesion that is 1 cm or more in 2 dimensions by CT scan
* Class A or B Child-Pugh liver classification
* No prior CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3*
* Platelet count at least 100,000/mm^3*
* Hemoglobin at least 8.5 g/dL* NOTE: *More than 7 days since prior blood transfusions or growth factors

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Albumin greater than 2.5 g/dL
* AST and ALT no greater than 3 times ULN
* INR no greater than 1.5 (unless receiving anticoagulants)

Renal

* Creatinine no greater than 2 times ULN

Cardiovascular

* LVEF at least 50%
* No New York Heart Association class III or IV cardiac disease
* No acute anginal symptoms

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study
* No severe concurrent disease, infection, or co-morbidity that would preclude study entry
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy for HCC
* No concurrent therapeutic biological response modifier

Chemotherapy

* No prior chemotherapy for HCC
* No prior chemoembolization for HCC
* No other concurrent cytotoxic chemotherapy

Endocrine therapy

* At least 6 weeks since prior hormonal therapy (an indicator lesion must exist outside the area of therapy
* No concurrent hormonal anticancer therapy

Radiotherapy

* No prior radiotherapy for HCC
* At least 6 weeks since prior radiofrequency ablation, selective internal radiation, or embolization (an indicator lesion must exist outside the area of therapy)
* No concurrent radiotherapy (including palliative therapy)

Surgery

* At least 6 weeks since prior surgical resection (an indicator lesion must exist outside the area of therapy)

  * Recurrence at the margin of the surgical resection is allowed
* At least 6 weeks since prior cryosurgery
* More than 4 weeks since other prior major surgery

Other

* More than 4 weeks since prior investigational therapy
* At least 6 weeks since prior intratumoral ethanol injection (an indicator lesion must exist outside the area of therapy)
* No other concurrent investigational anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-11; Primary Completion 2004-03 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna M. Brell, MD, Study Chair — Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center, Cleveland, Ohio, United States